CLINICAL TRIAL: NCT00059319
Title: Reduced Manipulation of the Aorta and Neurobehavioral Outcome Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: R01NS037242 (NIH)
Record Dates: First submitted 2003-04-23; First posted 2003-04-24 (Estimated); Last update posted 2007-05-21 (Estimated); Status verified 2007-05

CONDITIONS: Coronary Disease
Keywords: coronary artery bypass graft surgery; CABG surgery; neurobehavioral impairment; aorta clamping; aorta manipulation; microemboli
MeSH Terms: conditions — Coronary Disease

INTERVENTIONS:
Procedure: single aorta clamp with retrograde cardioplegia
Procedure: multiple aorta clamps with antegrade cardioplegia

SUMMARY:
The purpose of this trial is to determine whether aortic manipulation in patients undergoing coronary bypass graft surgery leads to increased incidence of microemboli and subsequent impairment of neurobehavioral function.

DETAILED DESCRIPTION:
Patients who have coronary artery bypass graft (CABG) surgery must have their aorta (the large blood vessel that is attached to the heart) clamped with an instrument. There are two basic ways of manipulating the aorta during surgery. One way is to place a single clamp across the aorta. The other way is to place more than one clamp on the aorta in several places. Both methods are used, but it is not known if one way is better than the other.

The purpose of this study is to compare the two methods of clamping to see if one way is better than the other, and to determine whether patients who undergo reduced manipulation of the aorta have fewer microemboli delivered to the brain during CABG surgery and have a lower incidence of neurobehavioral problems following surgery. Microemboli are tiny fat particles that enter the bloodstream during surgery, circulate to the brain, and block tiny blood vessels, causing brain deficits.

Participants in this trial will be randomly classified into one of two groups: the experimental group will undergo cross clamping of the aorta with a single clamp and be given retrograde cardioplegia for heart protection, and the control group will undergo cross clamping of the aorta with multiple clamps and be given antegrade cardioplegia for heart protection. Neurobehavioral assessments will be accomplished with a comprehensive battery of neurological and neuropsychological tests.

ELIGIBILITY:
* Participants must be English-speaking patients,
* 50 years of age or older, and
* undergoing elective CABG surgery.
* Participants of both genders and all races are eligible.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 1999-01

CONTACTS AND LOCATIONS:
Overall Officials: John W. Hammon, M.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States